CLINICAL TRIAL: NCT05223842
Title: Targeting Positive Emotions to Prevent Emotional Disturbances in Children During COVID-19
Brief Title: Family Promoting Positive Emotions Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Autumn Kujawa, Assistant Professor of Psychology and Human Development, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 211324
Record Dates: First submitted 2021-10-04; First posted 2022-02-04 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anhedonia; Stress; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorder; Mood Disturbance
Keywords: Depression; Anhedonia; Stress; Reward; Mental disorders; Mood disorders
MeSH Terms: conditions — Depression; Anhedonia; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Promoting Positive Emotions Group (Experimental): Each dyad (mother and their child) will receive 8 sessions of promoting positive emotions intervention with a clinician for 8 weeks.
  Interventions: Behavioral: Family Promoting Positive Emotions (F-PPE)
- Written Information Group (Active Comparator): Mothers will be sent written information and resources on depression for 8 weeks over email.
  Interventions: Behavioral: Written Information

INTERVENTIONS:
Behavioral: Family Promoting Positive Emotions (F-PPE) — F-PPE is an 8-session dyadic intervention designed to enhance positive emotionality and buffer against the effects of stress on anhedonia in children. The intervention will be administered online through videoconferencing sessions with a clinician to mothers and their children.
  Arms: Family Promoting Positive Emotions Group
Behavioral: Written Information — Mothers assigned to the Written Information condition will receive email newsletters providing resources relevant to depression.
  Arms: Written Information Group

SUMMARY:
Anhedonia is characterized by loss of interest or pleasure. The proposed pilot study would be the first to test an innovative, neuroscience-informed intervention in mothers reporting depressive symptoms and stress to enhance positive emotionality with the goal of preventing anhedonia and associated emotional disturbances in their children. This study will recruit dyads (mothers and their children) for the intervention.

DETAILED DESCRIPTION:
Anhedonia, characterized by loss of interest or pleasure, is a primary symptom of depression. Depression is increasingly prevalent and can cause significant impairments in life functioning. Given the increased presence of stress during COVID-19, there is a significant need for interventions that can prevent the development of anhedonia and depression. This study examines a neuroscience-informed positive emotion intervention to determine its effects on preventing anhedonia and associated emotional disturbances in dyads of children and their mothers. Participants will be randomized to either receive the positive emotion intervention for 8 sessions for 8 weeks with a clinician or the self-administered written information condition. Depressive symptoms, anhedonia, stress and other internalizing disorders will be assessed at baseline, and at the end of the intervention.

ELIGIBILITY:
Inclusion criteria for mothers:

* Age 18 and older who report at least subthreshold current depressive symptoms (> score of 8 on the Patient Health Questionnaire) and moderate COVID-19-related stress
* Can read and speak in English.
* Have access to a computer with a videoconferencing platform.

Inclusion criteria for children:

* Age 8-12 years who can participate with their biological mother who is 18 years or older that meets the above criteria.
* Can read and speak in English.

Exclusion criteria for mothers:

* Current substance use disorder.
* Intellectual disabilities.
* Diagnosis of mania or bipolar disorder.
* Diagnosis of a psychotic disorder (e.g., schizophrenia).
* Visual or hearing impairments that interfere with completing study measures and sessions.

Exclusion criteria for children:

* Diagnoses of autism spectrum disorders or developmental disorders.
* Intellectual disabilities.
* Diagnosis of mania or bipolar disorder.
* Diagnosis of a psychotic disorder (e.g., schizophrenia).
* Currently experiencing depressive symptoms.
* Visual or hearing impairments that interfere with completing study measures and sessions.
* Offspring of mothers who have previously participated in the study with another biological child.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Child perceived stress | 8 weeks
  The National Institutes of Health Toolbox Perceived Stress survey consists of 10 questions with options ranging in value from 1 to 5 to assess self-reported perceived stress for children (self- and parent-report). The minimum score is 10 and the maximum score is 50, with higher values meaning greater stress.
  Hypothesis 1a: Children in the F-PPE group will show lower post-intervention perceived stress compared to the written information group.
Child emotional distress | 8 weeks
  The Patient-Reported Outcomes Measurement Information System (Anxiety, Depression, Anger) short form consists of questions with five response options ranging in value from 1 to 5 to assess self-reported anxiety, depression, anger and irritability for participants (parent, child, and parent report). Total scores on the emotional distress scales for children range from 33 to 165 for self-report and 26 to 130 for parent report, with higher scores reflect greater distress.
  Hypothesis 1b: Children in the F-PPE group will show lower post-intervention emotional distress compared to the written information group.
Child positive affect | 8 weeks
  Positive affect will be assessed using the positive affect scale of the Positive and Negative Affect Schedule for Children administered through ecological momentary assessment over 10 days. Children rate their current affect on 5 items with a 1 to 5 scale for total scores from 5 to 25, with greater values reflecting greater positive affect.
  Hypothesis 2a: Children in the F-PPE group will show relative increases in daily positive affect from pre- to post-intervention compared to the written information condition.
  Hypothesis 2b: Changes in positive affect will partly account for F- PPE effects on child perceived stress and emotional distress.
  Hypothesis 2c: Changes in positive affect will partly account for F- PPE effects on child perceived stress and emotional distress.

SECONDARY OUTCOMES:
Child reward learning | 8 weeks
  Reward learning will be measured using a Reinforcement Learning Task. The extent to which children begin to preferentially select the button that is more likely to be reinforced as a reward across the task will be used to quantify reinforcement learning.
  Hypothesis 3a: Children in the F-PPE group will show relative increases in reward learning from pre- to post-intervention compared to the written information condition.
  Hypothesis 3b: Changes in reward learning will partly account for F- PPE effects on child perceived stress and emotional distress.
  Hypothesis 3c: Changes in reward learning will partly account for F- PPE effects on child perceived stress and emotional distress.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn J Kujawa, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available for sharing by request.
Time Frame: Immediately after publication.
Access Criteria: Principal investigator will review requests and grant access depending on the research question/plan and overlap with ongoing analyses in the laboratory.

REFERENCES:
- [Derived] Burkhouse KL, Dao A, Argiros A, Granros M, Cardenas E, Dickey L, Feurer C, Hill K, Pegg S, Venanzi L, Kujawa A. Targeting positive valence systems function in children of mothers with depressive symptoms: A pilot randomized trial of an RDoC-Informed preventive intervention. Behav Res Ther. 2023 Sep;168:104384. doi: 10.1016/j.brat.2023.104384. Epub 2023 Aug 9. PMID 37591042
- See also: Laboratory website — https://my.vanderbilt.edu/medlab/